CLINICAL TRIAL: NCT00468767
Title: A Phase III Prospective, Randomized, Double-Blind, Placebo-Controlled, Multi-Centred Tolerance and Efficacy Study of RSD1235 in Patients With Atrial Fibrillation
Brief Title: Phase III Tolerance and Efficacy Study of RSD1235 in Patients With Atrial Fibrillation
Acronym: ACT I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanz Pharma (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sheila Grant, VP of Product Development, Vernakalant, Cardiome Pharma Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1235-0703
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; RSD1235; Atrial fibrillation of 3 hours to 7 days duration.; Atrial fibrillation of 3 hours to 45 days duration.
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Atrial fibrillation (AF) duration of 3 hours to 7 days.
  Interventions: Drug: Vernakalant Injection 20 mg/mL
- 2 (Experimental): AF duration of >7 days to <45 days
  Interventions: Drug: Vernakalant Injection 20 mg/mL

INTERVENTIONS:
Drug: Vernakalant Injection 20 mg/mL
  Other Names: RSD1235; Vernakalant; Vernakalant Injection; Vernakalant (iv)

SUMMARY:
This study is being conducted to demonstrate the effectiveness of RSD1235 in the conversion of atrial fibrillation to sinus rhythm.

DETAILED DESCRIPTION:
There are approximately 2 million reported prevalent cases of atrial fibrillation (AF) and atrial flutter in the United States (Heart Disease & Stroke Statistics - 2003 Update, AHA). These arrhythmias may be occasional or sustained. While not directly fatal, these arrhythmias cause discomfort and can lead to stroke or congestive heart failure.

This Phase III trial is Cardiome's first pivotal study with RSD1235. The study seeks to confirm the findings of the Phase II proof-of-concept through demonstration of RSD1235's abilities to convert AF to sinus rhythm. The patient population will include recent onset AF (AF duration of 3 hours to 7 days) and patients with longer AF duration.

This is a double-blind, placebo-controlled, randomized study in patients with AF; stratification will be based on duration of AF. Treatment will be considered successful if there is a treatment-induced conversion of atrial arrhythmia to sinus rhythm for a minimum of 1-minute by Hour 1.5 (Time 0 = start of first infusion). All patients will be evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Have an atrial arrhythmia with symptoms that has been sustained for greater than 3 hours and up to 45 days.
* Have adequate anticoagulant therapy.

Exclusion Criteria:

* Have a QRS > 0.14 seconds unless patient has pacemaker or uncorrected QT > 0.440 seconds as measured on a 12-lead ECG.
* Have serious diseases/illnesses that could interfere with the conduct or validity of the study or compromise patient safety.
* Have received intravenous Class I or Class III antiarrhythmic drugs or intravenous amiodarone within 24 hours prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2003-08; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate the effectiveness of RSD1235 in the conversion of atrial fibrillation to sinus rhythm. | The proportion of patients with atrial fibrillation (AF) of 3 hours to 7 days duration who have treatment-induced conversion of AF to sinus rhythm for a minimum duration of one minute in the first 90 minutes after the first exposure to study treatment.

SECONDARY OUTCOMES:
To assess the safety of RSD1235 in this patient population. | The proportion of patients with AF of 3 hours to 45 days duration who have treatment-induced conversion of AF to sinus rhythm for a minimum duration of one minute in the first 90 minutes after the first exposure to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Grant, MBA, Study Director — Advanz Pharma
Locations (49):
- United States (11):
  - University of California, Los Angeles, California
  - Regional Cardiology Associates, Sacramento, California
  - Florida Heart Institute, Orlando, Florida
  - James Haley VA Hospital, Tampa, Florida
  - Cardiac Arrhythmia Service, Massachusetts General Hospital, Boston, Massachusetts
  - Thoracic and Cardiovascular Institute, Lansing, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - Main Line Health Heart Center, Wynnewood, Pennsylvania
  - Medical College of Virginia, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (12):
  - Heart Health Institute, Rockyview General Hospital, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Hamilton Health Sciences, Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospitals (Civic & General), Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Emergency Medicine Research Program, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM-Hotel-Dieu de Montreal, Montreal, Quebec
  - Institute de Cardiologie de Quebec, Hopital Laval, Ste Foy, Quebec
  - Centre Hospitalier LeGardeur, Terrebonne, Quebec
- Denmark (20):
  - Aalborg University, Aalborg
  - Århus Amtssygehus, Med. kardiologisk, Aarhus
  - Amager Hospital, Med. Center, Copenhagen
  - H:S Bispebjerg Hospital, Copenhagen
  - Helsingor Sygehus, Kardiovaskulært, Elsinore
  - Centralsygehuset Esbjerg Varde, Esbjerg
  - Fredericia Sygehus, Fredericia
  - Frederikssund Sygehus, Frederikssund
  - Glostrup Amtssygehus, Glostrup Municipality
  - Haderslev Sygehus, Kardiologisk Laboratorium, Haderslev
  - Gentofte Amtssygehus, Hellerup
  - Herlev Amtssygehus, Kardiologisk, Herlev
  - Hillerod Sygehus, Medicinsk, Hillerød
  - Sygehus Vendsyssel Hjorring, Hjørring
  - Holstebro centralsygehus, Holstebro
  - Horsens Sygehus, Horsens
  - Hvidovre Hospital, Kardiologisk, Hvidovre
  - Kolding Sygehus, Kardiologisk ambulatorium, Kolding
  - Roskilde Amts Sygehus Køge, Køge
  - Sygehus Fyn Svendborg, Svendborg
- Sweden (6):
  - Universitetssjukhuset MAS, Malmo
  - Universitetssjukhuset, Molndal, Mölndal
  - Universityetssjukhuset, Orebro, Örebro
  - Danderyds sjukhus, Stockholm
  - Akademiska Sjukhuset, Uppsala, Uppsala
  - Centrallasarettet, Vasteras, Västerås

REFERENCES:
- [Derived] Stiell IG, Dickinson G, Butterfield NN, Clement CM, Perry JJ, Vaillancourt C, Calder LA. Vernakalant hydrochloride: A novel atrial-selective agent for the cardioversion of recent-onset atrial fibrillation in the emergency department. Acad Emerg Med. 2010 Nov;17(11):1175-82. doi: 10.1111/j.1553-2712.2010.00915.x. PMID 21175515
- [Derived] Roy D, Pratt CM, Torp-Pedersen C, Wyse DG, Toft E, Juul-Moller S, Nielsen T, Rasmussen SL, Stiell IG, Coutu B, Ip JH, Pritchett EL, Camm AJ; Atrial Arrhythmia Conversion Trial Investigators. Vernakalant hydrochloride for rapid conversion of atrial fibrillation: a phase 3, randomized, placebo-controlled trial. Circulation. 2008 Mar 25;117(12):1518-25. doi: 10.1161/CIRCULATIONAHA.107.723866. Epub 2008 Mar 10. PMID 18332267